CLINICAL TRIAL: NCT06177977
Title: Ultracompact Hand-Held Swept-Source Optical Coherence Tomography (SS-HH-OCT) as a Novel Diagnostic Modality for Early-Onset Retinal Dystrophies (EORDs)
Brief Title: SS-HH-OCT as a Novel Diagnostic Modality for Early-Onset Retinal Dystrophies (EORDs)
Acronym: SS-HH-OCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00113941
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Retinal Dystrophies
Keywords: Retinal dystrophy; Inherited retinal dystrophy; Early onset retinal dystrophies (EORDS)
MeSH Terms: conditions — Retinal Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Group 1 - Progressive Inherited retinal dystrophy (IRD) (Active Comparator): 100 participants with progressive IRD; the most common IRD seen at Duke Clinics.
  Interventions: Device: SS-HH-OCT
- Group 2 - Non-progressive Inherited Retinal Dystrophy (IRD) (Active Comparator): 20 participants with non-progressive IRD (n=20), a subset of IRDs that are less frequently referred to Duke Clinics
  Interventions: Device: SS-HH-OCT
- Group 3 - Control participants (Active Comparator): 50 participants with normal retinal anatomy undergoing anesthesia for strabismus surgery as part of their clinically-indicated care.
  Interventions: Device: SS-HH-OCT

INTERVENTIONS:
Device: SS-HH-OCT — The investigational swept source OCT systems with handheld UC handpieces used in this study were developed at Duke University. OCT systems are non-contact, in-vivo optical imaging technology. The OCT system creates real-time, non-invasive images of ocular microstructure. OCT devices held above or in front of the eye while the sweeping infrared OCT beam scans across the retina. In contrast to the visible light used in clinical eye examinations, because infrared light is not visible, the participant is not disturbed by the light. OCT imaging allows the capture of hundreds of B-scan (cross-sectional) images in seconds. These B-scans are then stacked to create a volume; the stack may be summed up to create a retinal image. These retinal images are similar to images acquired during retinal photography except that they were captured with infrared light and provide depth information. Each volume and B-scan image can be viewed individually to measure and analyze ocular pathology.
  Other Names: Swept-source Handheld Ultracompact Optical Coherence Tomography (HH UC OCT)

SUMMARY:
The goal of this observational study is to utilize a novel imaging system designed for high-resolution retinal imaging of neonates, infants and children to identify the signs of photoreceptor development and degeneration in children with early-onset inherited retinal dystrophies (EORDs). Participants will have research imaging with SS-HH-OCT at the time of clinically-indicated eye examinations or procedures. The investigators aim to establish the basis for utilization of OCT imaging in earlier diagnosis and disease monitoring in children with EORDs. This work will set data reference standards and IRD endpoints that can be used in clinical trials.

DETAILED DESCRIPTION:
What photoreceptor degenerative changes take place in children with early-onset inherited retinal dystrophies, and how is photoreceptor development in this patient population affected by genetic defects?

Our novel investigational SS-HH-OCT system features high scanning speed, long laser wavelength, and an ergonomic light-weight handheld design. The investigators hypothesize that imaging with this system will enable us to characterize early-onset retinal dystrophies (EORD)-associated PDCs in young children. To this end, the investigators propose the following specific aims:

Specific Aim 1: Optimize and demonstrate reproducibility of SS-HH-OCT imaging protocols to visualize photoreceptor development and degeneration in children with and without EORDs.

Specific Aim 2: Use SS-HH-OCT parameters to characterize biomarkers of foveal photoreceptor development and degeneration in children with EORDs versus healthy controls.

A total of 80 participants will be enrolled in this study. Participants' age between 0 through 8 years (<9 years).

For children with EORD, successful completion of this study will result in 1) a framework for reproducible OCT imaging; 2) characterization of biomarkers of retinal degeneration; 3) establishment of reference data by genetic variants 4) insights into foveal development. Additionally, this study will set pilot data of structure-function data and timeline of photoreceptor degeneration for future NIH funded studies.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Participant's age is between 0 through 8 years (<9 years)
* Parent/legal guardian gives consents for the imaging study
* No ocular media opacities that could preclude imaging
* Refractive error equal or lower than 6 diopters

For EORD participants (Groups 1-2):

Meets clinical and molecular diagnosis of EORD (clinical determined by PI). Molecular diagnosis criteria:

* Autosomal dominant gene: One pathogenic or likely pathogenic variant that meets the clinical phenotype
* Autosomal recessive gene: two pathogenic or likely pathogenic variants in-trans which meet the phenotype.
* X-linked gene: one pathogenic or likely pathogenic variant which meets the phenotype.

For Controls (Group 3): No evidence of retinal pathology

Exclusion Criteria:

For all participants:

* Parent/legal guardian unwilling or unable to provide consent
* Refractive error higher than 6.00 diopters
* Participant has media opacities that preclude imaging
* Any non-IRD ocular condition that confound results interpretation such as glaucoma, uveitis, neurologic conditions affecting the optic nerve, etc.

For EORD participants (Groups 1-2): Does not meet molecular diagnosis criteria

For Controls (Group 3): Any suspicion of IRD

Ages: 0 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with abnormal microanatomy as measured by OCT reading | Up to 24 months
  Presence of abnormal retinal microanatomy as measured by OCT reading
Thickness of the participants retina at the fovea and surrounding optic nerve as measured by OCT reading | Up to 24 months
  Retinal thickness (microns) at the fovea and surrounding optic nerve

CONTACTS AND LOCATIONS:
Overall Officials: Ramiro Maldonado, MD, Principal Investigator — Duke University Eye Center
Locations (1):
- Duke University Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No